CLINICAL TRIAL: NCT00873002
Title: Phase I Study of Combination of Sorafenib and LBH589 in Hepatocellular Carcinoma
Brief Title: Panobinostat and Sorafenib in Treating Patients With Liver Cancer That is Metastatic and/or Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Dose Limiting Toxicity
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE6208; P30CA043703 (NIH); CASE6208 (Other: Case Comprehensive Cancer Center); CLBH589BUS23T
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; recurrent adult primary liver cancer; localized unresectable adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Panobinostat; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LBH589 (Active Comparator): This study utilizes a sequential dose-escalation design to define the MTD of LBH589 when combined with standard doses of sorafenib.
  Interventions: Drug: panobinostat; Drug: sorafenib tosylate

INTERVENTIONS:
Drug: panobinostat — Dose escalation: 7.5 mg/m2 day 1 and day 8 of 21 days cycle 10 mg/m2 day 1 and day 8 of 21 days cycle 15 mg/m2 day 1 and day 8 of 21 days cycle 20 mg/m2 day 1 and day 8 of 21 days cycle 30 mg/m2 day 1 and day 8 of 21 days cycle
Drug: sorafenib tosylate — 400 mg PO BID

SUMMARY:
RATIONALE: Panobinostat and sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Sorafenib may also stop the growth of liver cancer by blocking blood flow to the tumor.

PURPOSE: This phase I trial is studying the side effects and best dose of panobinostat when given together with sorafenib in treating patients with liver cancer that is metastatic and/or cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the safety and tolerability of panobinostat when combined with standard doses of sorafenib tosylate in patients with metastatic and/or unresectable hepatocellular carcinoma.
* Determine the maximum tolerated dose of panobinostat when combined with standard doses of sorafenib tosylate in these patients.

Secondary

* Determine the response rate.
* Determine the progression-free survival.
* Determine the overall survival rate.

OUTLINE: This is a dose escalation study of panobinostat.

Patients receive panobinostat IV on days 1 and 8 and oral sorafenib tosylate twice daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed for 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed hepatocellular carcinoma

  * Metastatic and/or unresectable disease
  * Child-Pugh score A or B

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Neutrophil count > 1500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (≤ 5.0 times ULN if elevation due to disease involvement)
* Serum bilirubin ≤ 1.5 times ULN
* Serum creatinine ≤ 1.5 times ULN or creatinine clearance ≥ 50 mL/min
* Total serum calcium (corrected for serum albumin) or ionized calcium ≥ lower limit of normal (LLN)
* Serum potassium ≥ LLN
* Serum sodium ≥ LLN
* Serum albumin ≥ LLN or 3 g/dL
* LVEF ≥ LLN as demonstrated by baseline MUGA or ECHO
* TSH and free T4 within normal limits (thyroid hormone replacement therapy allowed)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception (one being a barrier method) during and for 3 months after completion of study treatment
* INR < 1.5 or PT/PTT within normal limits
* No impaired cardiac function including any 1 of the following:

  * QTc > 450 msec on screening ECG
  * Congenital long QT syndrome
  * History of sustained ventricular tachycardia
  * History of ventricular fibrillation or torsades de pointes
  * Bradycardia, defined as heart rate < 50 beats per minute

    * Patients with a pacemaker and heart rate ≥ 50 beats per minute are eligible
  * Myocardial infarction or unstable angina within the past 6 months
  * Congestive heart failure (NYHA class III-IV)
  * Right bundle branch block and left anterior hemiblock (bifascicular block)
* No uncontrolled hypertension
* No thrombolic or embolic events (e.g., cerebrovascular accident and transient ischemic attacks) within the past 6 months
* No pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within the past 4 weeks
* No other hemorrhage/bleeding event > CTCAE Grade 3 within the past 4 weeks
* No unresolved diarrhea > CTCAE grade 1
* No other concurrent severe and/or uncontrolled medical conditions
* No other primary malignancy within the past 5 years except curatively treated carcinoma in situ of the cervix or basal cell or squamous cell carcinoma of the skin
* No serious non-healing wound, ulcer, or bone fracture
* No evidence or history of bleeding diathesis or coagulopathy
* No significant traumatic injury within the past 4 weeks
* No known or suspected allergy to sorafenib tosylate or any other study drug
* No condition that would impair a patient's ability to swallow whole pills
* No malabsorption problem
* No known human immunodeficiency virus (HIV) or hepatitis C positivity (baseline testing for HIV and hepatitis C is not required)
* No significant history of non-compliance to medical regimens

PRIOR CONCURRENT THERAPY:

* No prior HDAC inhibitors, DAC inhibitors, HSP90 inhibitors, sorafenib tosylate, or valproic acid for the treatment of cancer
* More than 4 weeks since prior chemotherapy, investigational drugs, or major surgery and recovered
* More than 4 weeks since open biopsy
* More than 5 days since prior and no concurrent valproic acid for any medical condition
* No concurrent St. John's wort or rifampin
* No concurrent drugs with a risk of causing torsades de pointes
* No concurrent CYP3A4 inhibitors
* No concurrent radiotherapy
* No concurrent grapefruit, grapefruit juice, or Seville (sour) oranges
* No other concurrent investigational therapy
* No other concurrent anticancer agents
* Concurrent anticoagulation treatment with warfarin or heparin allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-03; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Assessment of Safety and Tolerability | 6months to 1 year
  •Primary objective of the phase I trial will be to assess the safety and tolerability and to determine the maximum tolerated dose (MTD) of LBH 589 when combined with standard doses of sorafenib in the treatment of hepatocellular carcinoma.

SECONDARY OUTCOMES:
Progression-free survival | 6mo 1 year
  Evaluate time to progression vs progression free survival
Overall survival | until death
  Overall survival (OS) will be measured from study entry until death from any cause.
Response as assessed by RECIST | every 42 days
  To ensure comparability, baseline methods and on-study methods for response assessment must be performed using identical techniques. In addition, all subjects with evidence of objective tumor response (CR, PR or SD) should have the response confirmed with repeat assessments at least 21 days after the first documentation of response, resuming bimonthly (every 42 days) assessments thereafter. Objective tumor response will be assessed using the RECIST method.
Adverse events and abnormal laboratory value severity as assessed by NCI CTCAE version 3.0 | weekly during treatment to 30 days after treatment
  Events should be documented and recorded at each visit. Subjects should be followed for adverse events for 30 days after the last protocol related assessment, or until drug-related toxicities have resolved, whichever is later.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kim, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/show/NCT00873002?term=case6208&rank=1